CLINICAL TRIAL: NCT04998968
Title: Quality of Life in Patients With Permanent Hypoparathyroidism After Total Thyroidectomy in a Swedish Population Based Cohort
Brief Title: Quality in Patients With Permanent Hypoparathyroidism After Total Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01997
Record Dates: First submitted 2021-08-09; First posted 2021-08-10 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Permanent Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients with permanent hypoparathyroidism after total thyroidectomy: Patients with permanent hypoparathyroidism after total thyroidectomy for benign thyroid disease. These patients should be operated between 2005-2015 in Uppsala-Örebro healthcare region. Permanent hypoparathyroidism is defined as treatment with Calcium and/or vitamin D more than 12 months after surgery.
- Patients without permanent hypoparathyroidism after total thyroidectomy: Patients without permanent hypoparathyroidism after total thyroidectomy for benign thyroid disease. These patients should be operated between 2005-2015 in Uppsala-Örebro healthcare region.

SUMMARY:
Quality of life study. The study with include all patients operated with total thyroidectomy between 2005-2015 in Uppsala-Örebro healthcare region, Sweden. The study population has been identified in a previous study and includes close to 1700 patients, of which about 200 developed permanent hypoparathyroidism after surgery.

Quality of Life will be assessed using SF-36 Health Surgery and the outcome for patients with and without permanent hypoparathyroidism will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Total thyroidectomy between 2005-2015 in Uppsala-Orebro healthcare region.

Exclusion Criteria:

* Malignancy
* Sternotomy
* Previous thyroid surgery
* Previous or concurrent parathyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients are identified through the national quality registry for endocrine surgery, SQRTPA and the Swedish National Patient Register
Sampling Method: Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life using SF-36 short form | 2021
  The SF-36 yields eight scale scores and two summary scores, the physical component summary (PCS) and mental component summary (MCS). Scoring PCS and MCS involves three steps: 1) standardization of the scales (z-scores) 2) aggregation of score scales and 3) transformation of summary scores (t-scores). For each domain (PCS and MCS) the mean score is 50 with a standard deviation of 10. Higher scores indicates better quality of life (score range 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Olov Norlén, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No